CLINICAL TRIAL: NCT01768923
Title: Effect of Treat-to-target Strategies Aiming at Remission Compared With Minimal Disease Activity on Arterial Stiffness in Early Rheumatoid Arthritis - a Randomised Controlled Study
Brief Title: Early RA Vascular Randomised Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERA-Alx-2012
Record Dates: First submitted 2013-01-03; First posted 2013-01-16 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Early Rheumatoid Arthritis
Keywords: Early Rheumatoid Arthritis; Arterial stiffness; SDAI remission group; Minimal disease activity remission group
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SDAI remission group (Active Comparator): SDAI remission
  Interventions: Procedure: SDAI remission
- Minimal disease activity group (Active Comparator): Minimal disease activity remission
  Interventions: Procedure: Minimal disease activity remission

INTERVENTIONS:
Procedure: SDAI remission — SDAI remission group aims at the 2011 ACR/EILAR definition of remission (simplified disease activity score [SDAI] <3.3)
  Arms: SDAI remission group
Procedure: Minimal disease activity remission — Minimal disease activity group aims at minimal disease activity (DAS28<2.6) (minimal disease activity group)
  Arms: Minimal disease activity group

SUMMARY:
To investigate the effect of two tight-control treatment strategies, aiming at 1) 2011 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) definition of remission compare with 2) minimal disease activity (Disease Activity Index in 28 joints [DAS28] <2.6), on arterial stiffness in early rheumatoid arthritis (RA) patients.

To compare the effect of two treatments on arterial stiffness in Early Rheumatoid Arthritis

DETAILED DESCRIPTION:
One hundred RA patients with active disease (DAS28 >/=3.2), duration of symptoms less than 2 years, and are disease modifying anti-rheumatic drug naive will participate in this 5-year prospective, hospital-based, open-label, randomized, controlled trial.

All participants will receive 1-year tight-control treatment. One hundred patients will be randomly assigned to two arms. Treatment will be adjusted according to a standardized protocol every 3-monthly aiming at remission defined by the 2011 ACR/EULAR definition (Group 1, n=50, simplified disease activity score [SDAI] ≤3.3) or minimal disease activity (Group 2, n=50, DAS28<2.6). A follow up visit will be conducted at the 5th year to evulate long term effect on vascular outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* fulfilled the 2010 ACR/EULAR classification criteria for RA
* have symptoms onset of less than 2 years
* have active disease (DAS28> 3.2)
* are positive for rheumatoid factor or anti-cyclic citrullinated protein antibodies

Exclusion Criteria:

* have a history of overt cardiovascular diseases
* are on aspirin, or HMG-CoA reductase inhibitors (statins) or angiotensin-converting-enzyme inhibitor (ACEI)
* have severe renal impairment defined as a glomerular filtration rate of less than 30 ml/min/1.73m2
* have been previously treated with tumor necrosis factor alpha (TNFa) inhibitors or other biological DMARDs
* on glucocorticoids at a dose >10mg/day

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
The change in PWV over 1-year of treatment | Baseline and 12 months
  The change in PWV over 1-year of treatment

SECONDARY OUTCOMES:
The proportion of patients achieve clinical remission | 12 months
  The proportion of patients achieve clinical remission (SDAI</= 3.3 or DAS28<2.6) after 1-year treatment
The proportion of patients with a good response | 12 months
  According to EULAR definition, good response is DAS28 < 3.2 and a fall in score from baseline by > 1.2
ACR 20, 50, 70 responses | 12 months
  ACR 20, 50, 70 responses defined as at least 20%, 50%, 70% improvement in joint swelling and joint tenderness counts, and three of five other variables (i.e. ESR or CRP, HAQ score, pain score and physicians' and patients' global assessments)
The change in Alx@75 over 1-year of treatment | Baseline and 12 months
  Change in augmentation index over 1-year of treatment
The change in AIx@75 and PWV over 5-year of treatment | Baseline and 5-year
  long term effect on vascular outcomes (including changes in PWV and AIx) after 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Shan Tam, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Derived] Yue J, Wong PCH, Zhang Y, Peng F, Griffith JF, Xu J, Xiao F, Li TK, Hung V, Qin L, Tam LS. A novel visceral adiposity index predicts bone loss in female early rheumatoid arthritis patients detected by HR-pQCT. Sci Rep. 2023 Feb 11;13(1):2471. doi: 10.1038/s41598-023-29505-z. PMID 36774444
- [Derived] Tam LH, Shang Q, Li EK, Wong PC, Kwok KY, Kun EW, Yim IC, Lee VK, Yip RM, Pang SH, Lao VW, Mak QW, Cheng IT, Lau XS, Li TK, Zhu TY, Lee AP, Tam LS. Effect of Treat-to-target Strategies Aiming at Remission of Arterial Stiffness in Early Rheumatoid Arthritis: A Randomized Controlled Study. J Rheumatol. 2018 Aug;45(9):1229-1239. doi: 10.3899/jrheum.171128. Epub 2018 May 15. PMID 29764965